CLINICAL TRIAL: NCT03103971
Title: A Two-Stage Phase 1 Open-Label Study of huJCAR014, CD19-Targeted Chimeric Antigen Receptor (CAR)-Modified T Cells Bearing a Human Binding Domain, in Adult Patients With Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma and Acute Lymphocytic Leukemia
Brief Title: huJCAR014 CAR-T Cells in Treating Adult Patients With Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma or Acute Lymphoblastic Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to slow enrollment and end of funding
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Juno Therapeutics, Inc., a Bristol-Myers Squibb Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9364; NCI-2017-00421 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9364 (Other: Fred Hutch/University of Washington Cancer Consortium); RG9217000 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2017-03-27; First posted 2017-04-07 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent B-Cell Non-Hodgkin Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Primary Mediastinal (Thymic) Large B-Cell Lymphoma; Refractory Adult Acute Lymphoblastic Leukemia; Refractory B-Cell Non-Hodgkin Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory Primary Mediastinal (Thymic) Large B-Cell Lymphoma; Recurrent Transformed Non-Hodgkin Lymphoma; Recurrent High Grade B-Cell Lymphoma With MYC, BCL2, and BCL6 Rearrangements; Refractory High Grade B-Cell Lymphoma With MYC, BCL2, and BCL6 Rearrangements; Recurrent B Acute Lymphoblastic Leukemia; Recurrent Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Recurrent High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements; Refractory B Acute Lymphoblastic Leukemia; Refractory Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Refractory High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Burkitt Lymphoma | interventions — Cyclophosphamide; fludarabine; Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (leukapheresis, chemotherapy, huJCAR014) (Experimental): Patients undergo leukapheresis. Beginning 14-16 days after leukapheresis, patients undergo lymphodepleting chemotherapy comprising either cyclophosphamide IV daily for 1 day and fludarabine IV daily for 3 days or cyclophosphamide and fludarabine IV daily for 3 days. Within 36-96 hours after completion of lymphodepleting chemotherapy, patients receive huJCAR014 IV over 20-30 minutes on day 0.
  Interventions: Biological: Autologous Human Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing CD4+/CD8+ T-lymphocytes; Drug: Cyclophosphamide; Drug: Fludarabine; Other: Laboratory Biomarker Analysis; Procedure: Leukapheresis; Other: Pharmacological Study

INTERVENTIONS:
Biological: Autologous Human Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing CD4+/CD8+ T-lymphocytes — Given IV
  Other Names: Anti-CD19-CAR Genetically Engineered Autologous T Lymphocytes huJCAR014; Anti-CD19-CAR Genetically Engineered Autologous T-lymphocytes huJCAR014; Autologous Anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing CD4+/CD8+ T-lymphocytes; huJCAR014
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocytopheresis; Therapeutic Leukopheresis
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the side effects of huJCAR014 in treating patients with relapsed or refractory B-cell non-Hodgkin lymphoma or acute lymphoblastic leukemia. huJCAR014 CAR-T cells are made in the laboratory by genetically modifying a patient's T cells and may specifically kill cancer cells that have a molecule CD19 on their surfaces.

In Stage 1, dose-finding studies will be conducted in 3 cohorts:

1. Aggressive B cell NHL
2. Low burden ALL
3. High burden ALL

In Stage 2, studies may be conducted in one or more cohorts to collect further safety, PK, and efficacy information at the huJCAR014 dose level(s) selected in Stage 1 for the applicable cohort(s). There are two separate cohorts for stage 2:

1. Cohort 2A, CAR-naïve (n=10): patients who have never received CD19 CAR-T cell therapy.
2. Cohort 2B, CAR-exposed (n=27): patients who have previously failed CD19 CAR-T cell therapy.

DETAILED DESCRIPTION:
OUTLINE: This is a dose-escalation study of huJCAR014.

Patients undergo leukapheresis. Beginning 1-2 weeks after leukapheresis, patients undergo lymphodepleting chemotherapy comprising either cyclophosphamide intravenously (IV) daily for 1 day and fludarabine IV daily for 3 days or cyclophosphamide and fludarabine IV daily for 3 days. Alternative lymphodepleting chemotherapy regimens maybe used if patient's clinical situation or other logistical factors dictate otherwise. Within 36-96 hours after completion of lymphodepleting chemotherapy, patients receive huJCAR014 IV over 20-30 minutes on day 0.

After completion of study treatment, patients are followed up every 30 days for the first 3 months, every 3 months for up to 12 months, and then yearly for 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >= 18 years of age at the time of screening consent

INCLUSION CRITERIA FOR SCREENING

* Diagnosis of R/R B-cell NHL or ALL as defined below:

  * Relapsed or refractory B-cell NHL meeting all of the following criteria:

    * Diffuse large B-cell lymphoma (DLBCL), not otherwise specified (NOS); high grade B cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements; LBCL transformed from any indolent histology; or primary mediastinal B-cell lymphoma (PMBCL)
    * Prior treatment with an anthracycline and rituximab or another CD20-targeted agent (unless the disease is CD20-negative); transformed DLBCL (tDLBCL) must have failed treatment for DLBCL
    * At least one of the following:

      * Refractory disease after frontline chemo-immunotherapy
      * Not eligible for autologous hematopoietic stem cell transplant (auto-HSCT)
      * Relapsed or refractory disease after at least 2 lines of therapy or after auto-HSCT
      * Relapsed or refractory disease after allogeneic hematopoietic stem cell transplant (allo-HSCT)
  * Relapsed or refractory B-cell ALL (patients with Burkitt's lymphoma/leukemia are not eligible)
  * All B-ALL patients must have detectable disease by morphology, flow cytometry, cytogenetic analysis (e.g. polymerase chain reaction [PCR], fluorescence in situ hybridization [FISH], karyotyping) or imaging (e.g. positron emission tomography [PET]/computed tomography [CT]) or a high likelihood of active disease

    * Refractory: failure to achieve complete response (CR) (minimal residual disease [MRD]-negative) at the end of induction
    * Relapsed: recurrence of disease after achieving CR
* Evidence of CD19 expression by immunohistochemistry or flow cytometry on any prior or current tumor specimen or high likelihood of CD19 expression based on disease histology

INCLUSION CRITERIA FOR LEUKAPHERESIS AND PRE-THERAPY EVALUATION

* Screening evaluation appropriate for leukapheresis and T-cell collection
* Adequate vascular access available or planned for leukapheresis procedure (either peripheral line or surgically placed line)
* Documentation of CD19 expression on any prior or current tumor biopsy; patients who have received previous CD19-targeted therapy must have CD19-positive disease confirmed on a biopsy since completing the prior CD19-targeted therapy
* Internal review of histology
* Stage 2; cohort 2B (CAR-exposed) only:

  * Relapsed disease after achieving CR at the discretion of the principal investigator (PI) or designee, after prior CD19-targeted non-huJCAR014 CAR T-cell therapy. Patients who were in CR prior to the CD19-targeted non-huJCAR014 CAR T-cell therapy may be considered eligible at the discretion of the PI or designee. OR
  * Persistent disease after achieving PR at the discretion of the PI or designee, after prior CD19-targeted non-huJCAR014 CAR T-cell therapy. Patients who are less than 3 months from prior CD19-targeted non-huJCAR014 CAR T-cell therapy must have persistent disease on biopsy or imaging (e.g. PET-CT or CT) evidence of disease progression

INCLUSION CRITERIA FOR LYMPHODEPLETING CHEMOTHERAPY AND huJCAR014 TREATMENT

* Successful collection of T cells for huJCAR014 manufacturing
* Detectable disease by imaging (for example PET +/- CT, magnetic resonance imaging [MRI]) and/or pathology evaluation
* Karnofsky performance status >= 60%
* Assessed by the investigator to have adequate bone marrow function to receive lymphodepleting conditioning chemotherapy
* Serum creatinine =< 1.5 x age-adjusted upper limit of normal (ULN) or calculated creatinine clearance (Cockcroft and Gault) > 30 mL/min/1.73 m^2
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 5 x ULN and total bilirubin < 2.0 mg/dL unless due to malignancy or Gilbert's syndrome in the opinion of the PI or designee
* Common Terminology Criteria for Adverse Events (CTCAE) grade =< 1 dyspnea and oxygen saturation (SaO2) >= 92% on room air
* Left ventricular ejection fraction (LVEF) >= 40% as assessed by echocardiogram (ECHO) or multiple uptake gated acquisition (MUGA) scan performed within 1 month before starting lymphodepleting chemotherapy
* Women of childbearing potential (defined as all women physiologically capable of becoming pregnant) must agree to both of the following:

  * Use highly effective methods of contraception for at least 6 months after the last dose of huJCAR014, and
  * Have a negative serum pregnancy test performed within 28 days before starting lymphodepleting chemotherapy
* Males who have partners of childbearing potential must agree to use an effective barrier contraceptive method for at least 6 months after the last dose of huJCAR014

Exclusion Criteria:

EXCLUSION CRITERIA FOR SCREENING

* For patients in stage 1 only, prior treatment with any CD19 CAR T-cell therapy is excluded
* Known active hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) infection
* Pregnant or breastfeeding women
* Any known contraindication to leukapheresis
* Any known and irreversible contraindication to huJCAR014 therapy
* Medical, psychological, familial, sociological, or geographical condition that does not permit compliance with the protocol as judged by the PI or designee, or unwillingness or inability to follow protocol procedures

EXCLUSION CRITERIA FOR LEUKAPHERESIS AND PRE-THERAPY EVALUATION

* History or presence of clinically relevant central nervous system (CNS) pathology that, in the opinion of the PI or designee, is a contraindication to lymphodepleting chemotherapy or huJCAR014 infusion
* History of another primary malignancy that has not been in remission for at least 2 years with the following exceptions: nonmelanoma skin cancer, curatively treated localized prostate cancer, cervical carcinoma in situ on biopsy or a squamous intraepithelial lesion on Pap smear, or other malignancy considered by the investigator to have a low risk of relapse or progression
* Active autoimmune disease requiring immunosuppressive therapy, unless considered by the PI or designee to be eligible
* Presence of active acute or chronic graft versus host disease (GVHD)
* Use of any of the following:

  * Cytotoxic or lymphotoxic agents (including prednisone > 5 mg/day or equivalent corticosteroid) within 1 week prior to leukapheresis; physiologic corticosteroid replacement, and topical or inhaled corticosteroids are not excluded
  * GVHD therapies within 4 weeks prior to leukapheresis (e.g., calcineurin inhibitors, methotrexate or other chemotherapeutics, mycophenolate, rapamycin, thalidomide, immunosuppressive antibodies such as anti-TNF, anti-IL-6, or anti-IL-6R)
  * Experimental agents within 4 weeks prior to leukapheresis unless progression is documented on therapy and at least 3 half-lives have elapsed prior to leukapheresis
  * Radiation encompassing all sites of known tumor within 6 weeks prior to leukapheresis, unless there is evidence of active disease after radiation by imaging, biopsy or clinical evaluation
  * Allo-HSCT within 60 days prior to leukapheresis or donor lymphocyte infusion (DLI) within 6 weeks prior to leukapheresis
  * Treatment with cladribine within 3 months prior to leukapheresis
  * Treatment with alemtuzumab within 3 months prior to leukapheresis

EXCLUSION CRITERIA FOR LYMPHODEPLETING CHEMOTHERAPY AND huJCAR014 TREATMENT

* Uncontrolled and serious infection
* Presence of active acute or chronic GVHD
* DLI within 6 weeks prior to lymphodepletion chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2024-03-23 (Actual)

PRIMARY OUTCOMES:
Incidence of toxicity | Up to 30 days after the final dose of study therapy
  Will be graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. All adverse events (AEs) will be listed and summarized. Summaries of laboratory data will include, at a minimum, treatment-emergent laboratory abnormalities. Summaries of AEs and laboratory abnormalities will be based on the All Treated analysis set.
Dose-limiting toxicity (DLT) rates | Up to 28 days
  Observed DLT rates will be summarized based on the DLT-Evaluable analysis set. Final DLT rates at each dose level will be estimated by isotonic regression.
Maximum concentration (Cmax) of autologous human anti-CD19CAR-4-1BB-CD3zeta-EGFRt-expressing CD4+/CD8+ T-lymphocytes (huJCAR014) cells in blood | Up to 28 days
  huJCAR014 will be measured in blood using quantitative polymerase chain reaction (PCR) (qPCR) and flow cytometry over 28 days after huJCAR014 infusion. Cmax is the peak concentration of huJCAR014 cells in blood in the first 28 days after infusion.
Time to maximum concentration (Tmax), of huJCAR014 cells in blood | Up to 28 days
  huJCAR014 will be measured in blood using quantitative PCR (qPCR) and flow cytometry over 28 days after huJCAR014 infusion. Tmax is the time to reach the maximum concentration of huJCAR014 cells in blood in the first 28 days.
Area under the curve of huJCAR014 cells in blood | Up to 28 days
  huJCAR014 will be measured in blood using quantitative PCR (qPCR) and flow cytometry over 28 days after huJCAR014 infusion. AUC is the calculated area under the curve of huJCAR014 concentrations in blood by time after infusion through 28 days.
Presence of huJCAR014 cells in bone marrow | Up to 28 days
  The persistence of huJCAR014 in the bone marrow at 28 days will be assessed, based on both a qPCR assay and flow cytometry.

SECONDARY OUTCOMES:
Complete response (CR) rate | Up to 15 years
  Will be summarized along with the 2-sided 95% exact Clopper-Pearson confidence intervals based on the efficacy-evaluable (EE) analysis sets. In addition, CR rate will be presented based on the all-treated analysis set
Partial response (PR) rate | Up to 15 years
  Will be summarized along with the 2-sided 95% exact Clopper-Pearson confidence intervals based on the EE analysis sets.
Objective response rate (ORR) | Up to 15 years
  Will be defined as the proportion of patients with a best response of either CR or PR. Will be summarized along with the 2-sided 95% exact Clopper-Pearson confidence intervals based on the EE analysis sets. In addition, ORR will be presented based on the All-Treated analysis set.
Duration of response (DOR) | Up to 15 years
  Will be defined as the time from date of first response to relapse/progression or death. Kaplan-Meier (KM) methodology will be used to analyze DOR.
Progression-free survival (PFS) | From date of first huJCAR014 infusion to progressive disease or death, assessed up to 15 years
  KM methodology will be used to analyze PFS.
Event-free survival (EFS) | From the date of the first huJCAR014 infusion to death from any cause, relapse, or treatment failure, whichever occurs first, assessed up to 15 years
  KM methodology will be used to analyze EFS.
Overall survival (OS) | From date of first huJCAR014 infusion to death, assessed up to 15 years
  KM methodology will be used to analyze OS.

OTHER OUTCOMES:
Cellular immune responses to huJCAR014 | Up to 1 year
  Percentage of patients with cellular immune responses to huJCAR014.
B-cell depletion in circulation | Up to 1 year
  Percentage of patients with B cells < 0.01% in blood.
Cytokine profile | Up to 1 year
  Peak concentration of IL-6 in blood after CAR-T cell infusion.
CD19 expression on tumor cells in biopsies | Up to 1 year
  Percentage of patients with CD19-negative disease after CAR-T cell infusion.
Phenotype of CAR T cells in blood | Up to 1 year
  Percentage of patients with CAR-T cells expressing CD62L.
Product attributes (e.g., cell phenotype, cytokine profiles) | Up to 1 year
  Product attributes (e.g., cell phenotype, cytokine profiles) will be correlated with AEs, pharmacokinetic (PK), and tumor response rates.
Tumor attributes (e.g., checkpoint expression) | Up to 1 year
  Tumor attributes (e.g., checkpoint expression) on PK will be correlated with biomarkers (e.g., peripheral cytokines).

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Gauthier, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gauthier J, Liang EC, Huang JJ, Kimble EL, Hirayama AV, Fiorenza S, Voutsinas JM, Wu QV, Jaeger-Ruckstuhl CA, Pender BS, Kirchmeier DR, Torkelson A, Braathen K, Basom R, Shadman M, Kopmar NE, Cassaday RD, Riddell SR, Maloney DG, Turtle CJ. Phase 1 study of CD19 CAR T-cell therapy harboring a fully human scFv in CAR-naive adult patients with B-ALL. Blood Adv. 2025 Apr 22;9(8):1861-1872. doi: 10.1182/bloodadvances.2024015314. PMID 39820359